CLINICAL TRIAL: NCT03736668
Title: Study of Left Ventricular Function of Patients With Type 2 Diabetes Without Cardiovascular Disease
Acronym: DIACAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DIACAR
Record Dates: First submitted 2018-10-31; First posted 2018-11-09 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Type2 Diabetes
MeSH Terms: interventions — Echocardiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Type 2 diabetes (Experimental): One year after patient's inclusion, during the additional cardiology consultation, an echocardiography will be performed by the investigator to evaluate any changes.
  Two years after the patient's inclusion, an investigator will contact by phone the general practitioner, cardiologist and / or diabetologist treating the patient to find out if any cardiovascular events occurred.
  Interventions: Diagnostic Test: echocardiography

INTERVENTIONS:
Diagnostic Test: echocardiography — One year after patient's inclusion, an echocardiography / doppler will be performed to evaluate any changes.Two years after the patient's inclusion, an investigating cardiologist will contact the physician, cardiologist and / or diabetologist treating the patient by telephone to find out if any cardiovascular events have occurred.

SUMMARY:
Type 2 diabetes is associated with high cardiovascular risk. Recent meta-analyzes suggest that the risk of hospitalization for heart failure in the diabetic is increased by 20% for each hemoglobin A1c point and that the risk of death from all causes or cardiovascular cause and the risk of hospitalization is significantly increased by 30 to 40% in patients with acute or chronic heart failure with diabetes.

Systematic analysis of cardiac function is not currently proposed in international recommendations even though some antidiabetic drugs have been associated with an increased risk of heart failure in large randomized controlled trials or an increase in adverse events in proof-of-concept studies of heart failure with or without diabetes. Observational studies suggest that hypoglycemic sulfonamides may increase the risk of developing heart failure. In contrast, two sodium-glucose cotransporter type 2 inhibitors (empagliflozin and canagliflozin) have recently demonstrated a significant reduction in hospitalizations for heart failure in two large randomized controlled trials.

The detection of subclinical left ventricular dysfunction is therefore essential to better assess the risk of cardiac decompensation and to identify the existence of possible contraindications to the use of certain classes of drugs used in diabetes. Recent studies suggest that the left ventricular ejection fraction measured on three-dimensional acquisitions is a prognostic value index greater than the ejection fraction measured by Simpson biplane method in two-dimensional ultrasound. Similarly, it seems that the analysis of global longitudinal deformation is a prognostic factor superior to the analysis of the ejection fraction (two-dimensional or three-dimensional). The investigators will analyze these different parameters to confirm these data.

DETAILED DESCRIPTION:
The main objective of this study is to analyze left ventricular function by echocardiography in a prospective cohort of 200 patients with type 2 diabetes and without known cardiac dysfunction and to search for possible differences in clinical profile depending on the presence and type of cardiac function's impairment.

Patients will be classified into four categories according to the left ventricular function:

* Normal heart function
* Altered ejection fraction (<40%)
* Ejection fraction preserved (> 50%) with structural abnormality (left ventricular hypertrophy, left atrial dilatation) or diastolic dysfunction
* Moderately impaired ejection fraction "mid range" (40 to 49%)

ELIGIBILITY:
Inclusion Criteria:

* Patient with age > 18 years
* Patient with type 2 diabetes with no history of proven cardiovascular disease
* Patient hospitalizes In Diabetes Week Hospital (HDS)
* Patient affiliated with a health insurance plan
* Patient able to give free, informed and express consent

Exclusion Criteria:

1. Patient with proven cardiovascular disease:

   * Acute coronary syndrome, revascularization of the myocardium, known and / or treated ischemic heart disease
   * Rhythmic disorders such as atrial fibrillation
   * Significant valvular disease known or treated by prosthetic valve
   * known and treated heart failure
   * Stroke
   * Symptomatic and / or revascularized arteritis
   * Pacemaker wearers
   * Cardiac Defibrillator Carriers
2. Patient with progressive cancer
3. Patient who has been treated with cardio-toxic chemotherapy or mediastinal radiotherapy
4. Patient under tutorship / curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2019-07-23 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Measurement of left ventricular ejection fraction | year 1
  During the electrocardiography, the left ventricular function will be measured to look for possible differences depending on the type of impairment of cardiac function. Patients will be classified into 4 categories: normal cardiac function, altered ejection fraction (<40%), preserved ejection fraction (>50%) with structural abnormality or diastolic dysfunction, or ejection fraction mid range (40 to 49%).

SECONDARY OUTCOMES:
Evaluation of the modification of left ventricular function | year 1
  During the electrocardiography, the left ventricular ejection fraction will be measured to look for possible differences depending on the type of impairment of cardiac function. Patients will be classified into 4 categories: normal cardiac function, altered ejection fraction (<40%), preserved ejection fraction (>50%) with structural abnormality or diastolic dysfunction, or ejection fraction mid range (40 to 49%).
Occurrence of major or fatal events, or cardiovascular events | year 1
  The investigator will collect major or fatal events, or cardiovascular events.
Occurrence of major fatal or cardiovascular events | year 2
  The investigator will contact by phone patient's general practitioner, cardiologist or diabetologist to collect major or fatal events, or cardiovascular events.
Comparison of left ventricular ejection fraction measurements performed by biplane Simpson with those obtained from a 3D acquisition (Philips HeartModel). | year 1
  During the electrocardiography, the left ventricular ejection fraction will be measured by biplane Simpson and a 3D acquisition. Then, the measurements will be compare.
Comparison of inter- and intra-observer variability in a sample of 20 patients in the cohort of 200 patients | Year 1
  The mesaurement of left ventricular function will be compare in in a sample of 20 patients in the cohort of 200 patients between operators.
Comparing the volume of the left atrium in Simpson biplane and in 3D | Year 1
  During the echocardiography, the volume of the left atrium will be measure in Simpson biplane and in 3D and then the measurements will be compare.

CONTACTS AND LOCATIONS:
Overall Officials: Yara P ANTAKLY, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France